CLINICAL TRIAL: NCT01487356
Title: Factors Associated With Short Withdrawal Time and Polyp Detection Rate During Colonoscopy
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H10-00312
Record Dates: First submitted 2011-08-03; First posted 2011-12-07 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-12

CONDITIONS: Colon Polyps
Keywords: Colonoscopy; quality assurance; withdrawal time; polyp detection rate
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing colonoscopy: Data was collected on all adult patients undergoing outpatient colonoscopy at St. Paul's Hospital from May 2008 to June 2009. Exclusion criteria were prior colon resection and repeat colonoscopy for the purpose of endoscopic therapy for known lesions.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Colonoscopies were conducted as per the endoscopist's usual practice. No change in protocol was expected.

SUMMARY:
Colonoscopy withdrawal times are a critical element in determining quality of colonoscopy; however, few studies have evaluated specific factors that may influence the duration of withdrawal, and specifically short withdrawal times. Other factors affecting polyp detection rate, one element of quality of colonoscopy, also need further study. By collecting data on hundreds of colonoscopies performed by 9 endoscopists, our goal was to identify factors associated with withdrawal time, inappropriately short withdrawal times, and polyp detection rate during colonoscopy.

DETAILED DESCRIPTION:
Background:

Colonoscopy withdrawal times are a critical element in determining quality of colonoscopy; however, few studies have evaluated specific factors that may influence the duration of withdrawal, and specifically short withdrawal times. Other factors affecting polyp detection rate, one element of quality of colonoscopy, also need further study.

Objective:

To identify factors associated with withdrawal time, inappropriately short withdrawal times, and polyp detection rate during colonoscopy.

Design:

Data were prospectively collected (05/08-06/09) on 802 colonoscopies conducted by 9 blinded endoscopists, including patient age and sex, indication, colonoscope insertion and withdrawal time, biopsies performed, number/size of polyps and method of resection, bowel preparation quality, time of day, day of week, endoscopist, position of the procedure within the endoscopist's slate, and call status of the endoscopist.

Setting:

This study was conducted at a single tertiary care hospital, St. Paul's Hospital, in Vancouver, British Columbia.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients undergoing colonoscopy at St. Paul's Hospital in Vancouver, BC.

Exclusion Criteria:

* Exclusion criteria were prior colon resection and repeat colonoscopy for the purpose of endoscopic therapy for known lesions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All adult patients undergoing colonoscopy at St. Paul's Hospital in Vancouver, BC.
Sampling Method: Non-Probability Sample
Enrollment: 802 (Actual)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rob Enns, MD, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada